CLINICAL TRIAL: NCT06022107
Title: Piloting a Novel Social Support Intervention for Addiction Recovery
Brief Title: Social Support Intervention for Addiction Recovery
Acronym: LDART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Society of Addiction Psychology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000035434; 000 (Other: CTGTY)
Record Dates: First submitted 2023-08-23; First posted 2023-09-01 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Alcohol; Harmful Use; Alcohol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- LDART (Experimental): Participants will be asked to log onto the LDART website each night for a month.
  Interventions: Behavioral: LDART

INTERVENTIONS:
Behavioral: LDART — LDART is a newly developed web-based social support intervention that can be accessed by smartphone or computer. Each night, the participant sets a recovery goal for the next day (e.g., drink less than usual, go to a support group meeting). The next night, they log on to LDART to indicate whether they reached their goal for the day. Depending on their response, they will be shown either a celebratory or encouraging message from someone in the addiction recovery community, along with specific information on that person's recovery organization.

SUMMARY:
The purpose of this research study is to determine whether using a web-based intervention is feasible, acceptable, and helpful for people who engage in hazardous alcohol use and want to cut down or quit.

DETAILED DESCRIPTION:
This pilot study will determine the feasibility and acceptability of a novel online social support intervention (Let's Do Addiction Recovery Together!, abbreviated as LDART) that uses pre-recorded videos created by members of recovery support services to help individuals in early recovery from hazardous alcohol use sustain motivation during recovery and introduce them to freely available recovery support services in the community. The investigators will recruit participants to use the web-based intervention daily for a month; they will also fill in questionnaires about their substance use and engagement with recovery support services at the beginning and end of the study to determine preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Is at the time of study participation residing in Connecticut, USA
* Is fluent in English and has a 6th grade reading level or higher
* Alcohol Use Disorders Identification Test (AUDIT) score of ≥8
* Has had at least one heavy drinking day in the past month
* Has some desire to cut down or quit their alcohol use
* Has a smartphone or computer with access to internet

Exclusion Criteria:

* Has vulnerable population status (e.g., pregnant people, prisoners)
* Is at the time of study participation receiving in-patient psychiatric treatment involving hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc N Potenza, MD, PhD, Principal Investigator — Yale University; Li Yan McCurdy, PhD, Principal Investigator — Yale University
Locations (1):
- 1 Church St, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCurdy LY, Kong G, Krishnan-Sarin S, Kiluk BD, Potenza MN. A non-randomized pilot study protocol of a novel social support intervention for individuals in early recovery from hazardous alcohol use. PLoS One. 2023 Oct 5;18(10):e0292293. doi: 10.1371/journal.pone.0292293. eCollection 2023. PMID 37796784

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LDART
Started | 30
Completed | 23
Not Completed | 7
Not completed — Did not complete baseline questionnaire / did not begin using intervention | 4
Not completed — Dropped out of study for higher level of care | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Of the 30 participants who were enrolled in the trial, 4 did not complete the baseline assessments and thus did not begin using the intervention.
Arm/Group | LDART
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Past-year AUDIT score [Mean (Standard Deviation); unit: units on a scale] — Alcohol Use Disorder Identification Test (AUDIT) is a screening tool for hazardous alcohol use. Range of score is from 0-40, where higher scores indicate greater severity. A score of ≥8 indicates hazardous alcohol use.
  units on a scale | 22.7 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility
Description: Feasibility of recruitment is measured as the number of adults who consent to study participation divided by the number of months the trial recruits for.
Time Frame: Baseline
Measure: Number; unit: participants per month
Arm/Group | LDART
Number analyzed (Participants) | 30
participants per month | 10

2. Primary Outcome: Retention Feasibility
Description: Retention rate is calculated as the number of participants who complete the study divided by the number of participants who consented to participating in the study.
Time Frame: One-month post-intervention (Day 56)
Population: Retention feasibility was calculated as the number of participants who completed the study (i.e., completed the one-month post-intervention assessment) divided by the number of participants who enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | LDART
Number analyzed (Participants) | 30
Participants | 23

3. Primary Outcome: Intervention Acceptability (Engagement With Intervention)
Description: Acceptability is calculated as the number of nights participants login to LDART within the 28-day window.
Time Frame: Duration of intervention (Days 1-28)
Population: The one participants who dropped out mid-intervention for higher level of care was excluded from analysis.
Measure: Mean (Standard Deviation); unit: nights
Arm/Group | LDART
Number analyzed (Participants) | 25
nights | 22.9 (4.3)

4. Primary Outcome: Intervention Acceptability (Subjective Experience)
Description: Acceptability is measured with a 9-item self-report acceptability assessment questionnaire. This comprises questions regarding the motivational and supportive properties of the content, perceptions on the frequency of engaging with the intervention, and whether they enjoyed using the intervention. Each question is rated on a 5-point Likert scale, where higher values indicate greater acceptability. There will also be two open-ended questions for participants to indicate what they liked and did not like about the intervention and ways to improve it. Data reported here reflects percentage of participants who answered "agree" or "strongly agree" to the question: "I would recommend LDART to someone trying to cut down or quit drinking".
Time Frame: Post-intervention (Day 28)
Population: Of the 25 participants who completed the intervention, 3 did not complete the acceptability ratings, and 1 participant skipped this question.
Measure: Count of Participants; unit: Participants
Arm/Group | LDART
Number analyzed (Participants) | 21
Participants | 18

5. Secondary Outcome: Percentage of Drinking Days Per Month
Description: Timeline Follow Back is a validated, self-reported instrument that provides specific dates for alcohol use in the past 28 days, and the number of standard drinks consumed on each drinking day. Percent Drinking Days Per Month is calculated as the percentage of days in the 28-day window in which one or more standard drinks is consumed for two consecutive windows.
Time Frame: Day 0 (Pre-intervention), 28 (Post-intervention), and 56 (1-month post-intervention)
Population: 2 of the 25 participants did not have data at the third time point (one month post-intervention) so were excluded from analyses.
Measure: Mean (Standard Deviation); unit: Percentage of days in a month
Arm/Group | LDART
Number analyzed (Participants) | 23
Percentage of days in a month
  Pre-intervention | 61.3 (31.2)
  During intervention | 45.2 (34.6)
  Post-intervention | 42.6 (34.2)

6. Secondary Outcome: Percentage of Heavy Drinking Days Per Month
Description: Percent Heavy Drinking Days is calculated from the Timeline Follow Back instrument as the number of days in the 28-day window in which four/five or more standard drinks is consumed for women/men for two consecutive windows.
Time Frame: Day 0 (Pre-intervention), 28 (Post-intervention), and 56 (1-month post-intervention)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of days in a month
Arm/Group | LDART
Number analyzed (Participants) | 23
Percentage of days in a month
  Pre-intervention | 27.1 (30.0)
  During intervention | 17.1 (22.5)
  Post-intervention | 17.9 (23.2)

7. Secondary Outcome: Hours Spent Engaging With Recovery Support Services
Description: Self-reported total number of hours spent engaging in recovery support services (e.g., being at a recovery community center, attending a support group meeting) in the past 28-day time window for two consecutive windows.
Time Frame: Day 0 (Pre-intervention), 28 (Post-intervention), and 56 (1-month post-intervention)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours in a month
Arm/Group | LDART
Number analyzed (Participants) | 23
hours in a month
  Pre-intervention | 2.4 (5.5)
  During intervention | 10.8 (25.4)
  Post-intervention | 7.6 (12.7)

8. Secondary Outcome: World Health Organization Quality of Life - Brief Version
Description: World Health Organization Quality of Life - Brief Version (WHOQOL-BREF) is a questionnaire with 24 items that correspond to four domains: physical health, psychological health, social relationships, and environment. Each question is rated on a five-point Likert scale. Each domain score is transformed based on the lowest possible score to create a modified range of 0-100 for each domain. All four domain scores are then averaged to create a single score on a range of 0-100, where higher values indicate higher quality of life.
Time Frame: Day 0 (Pre-intervention), 28 (Post-intervention), and 56 (1-month post-intervention)
Population: 2 of the 25 participants did not have data at the second time point (post-intervention); 1 of the 25 participants did not have data at the third time point (one month post-intervention), and 1 of the participants did not have data at either the second or third time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LDART
Number analyzed (Participants) | 21
score on a scale
  Pre-intervention | 57.1 (4.3)
  Post-intervention | 60.7 (4.4)
  1-month post-intervention | 60.1 (4.7)

9. Secondary Outcome: Brief Assessment of Recovery Capital
Description: Brief Assessment of Recovery Capital (BARC) is a 10-item self-report measure of recovery capital with ten domains (substance use and sobriety, global psychological health, global physical health, citizenship and community involvement, social support, meaningful activities, housing and safety, risk-taking, coping and life functioning, recovery experience). Total score ranges from 0-50, where higher values indicate higher recovery capital.
Time Frame: Day 0 (Pre-intervention), 28 (Post-intervention), and 56 (1-month post-intervention)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LDART
Number analyzed (Participants) | 21
score on a scale
  Pre-intervention | 43.9 (8.0)
  Post intervention | 46.9 (9.2)
  1-month post-intervention | 45.3 (7.9)

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | LDART
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT06022107/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT06022107/ICF_001.pdf